CLINICAL TRIAL: NCT01274767
Title: Prevention of Recurrent Ulcer Bleeding in High-risk Aspirin Users Who Are Not Infected With Helicobacter Pylori: A Prospective Cohort Study (NSAID#3NANC Study)
Brief Title: Prevention of Recurrent Ulcer Bleeding in High-risk Aspirin Users Who Are Not Infected With Helicobacter Pylori
Acronym: 3NANC
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Francis KL Chan, Professor, Chinese University of Hong Kong
Other Study IDs: 3NANC
Record Dates: First submitted 2011-01-11; First posted 2011-01-12 (Estimated); Last update posted 2017-04-24 (Actual); Status verified 2017-04

CONDITIONS: Ulcer Bleeding

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- High risk cohort: Patients having history of endoscopically confirmed ulcer bleeding, need long-term aspirin for cardiovascular or cerebrovascular prophylaxis and have a negative test for H. pylori based on histology
- Average risk cohort: Patients having no history of endoscopically confirmed ulcer bleeding, need long-term aspirin for cardiovascular or cerebrovascular prophylaxis and have H. pylori positive OR negative

SUMMARY:
Low-dose aspirin is the mainstay of treatment for patients with coronary heart disease and stroke. However, low-dose aspirin increases the risk of ulcer bleeding. Current evidence indicates that 80 - 100 mg of aspirin daily provides good protection against vascular events and the risk of ulcer bleeding is low (about 1% per year). Since the overall risk of bleeding is low, aspirin users who do not have previous ulcer disease do not require prophylaxis with anti-ulcer drugs. In contrast, aspirin users with a history of ulcer disease have a 2- to 4-fold increased risk of ulcer bleeding. The best strategy for reducing the risk of bleeding in high-risk aspirin users remains unclear. Current strategies for high-risk patients include the use of anti-ulcer drugs, elimination of risk factors (e.g. Helicobacter pylori), or the use of enteric-coated aspirin.

Although co-therapy of aspirin with an acid suppressant reduces the risk of ulcer bleeding, drug compliance may limit its clinical usefulness particularly in patients who are already receiving multiple drugs. The efficacy of enteric-coated aspirin in preventing ulcer complications showed conflicting results. One study found that enteric-coated aspirin increases the risk of ulcer bleeding. A recent study showed that enteric-coated aspirin causes minimal acute gastric injury.

The investigators postulated that among patients without H. pylori infection and a history of ulcer bleeding who continue to use low-dose aspirin, enteric-coated aspirin reduces the long-term risk of ulcer complications to a level that is comparable to that of average-risk aspirin users.

DETAILED DESCRIPTION:
Low-dose aspirin is increasingly used for the prophylaxis against coronary heart disease and stroke. However, it is also an important cause of peptic ulcer bleeding worldwide. In England and Wales, low-dose aspirin is estimated to account for about 10% of ulcer bleeding in people aged 60 and over [Weil 1995]. The problem of aspirin-related ulcer disease is expanding with the increasing use of aspirin for cardiovascular prophylaxis.

No dose of aspirin is entirely free of risk. Using a daily dose of aspirin as low as 75 mg, the risk of ulcer bleeding doubles that of non-users [Weil 1995]. Previous ulcer disease and concurrent major medical illnesses are important risk factors for ulcer bleeding with low-dose aspirin. Among aspirin users, those with previous ulcer disease have a 5-fold increased risk of ulcer bleeding [Lanas 2000].

Various strategies have been used to prevent recurrent ulcer bleeding in high-risk aspirin users, such as eradication of Helicobacter pylori, the use of prophylactic anti-ulcer drugs or enteric-coated aspirin. Recently, the investigators have shown that the eradication of H. pylori is comparable to maintenance treatment with omeprazole, a potent acid suppressant, in preventing recurrent ulcer bleeding for high-risk aspirin users [Chan 2001]. However, about 50% of aspirin users are not infected with H. pylori.

The optimal strategy to prevent ulcer complications for high-risk aspirin users who are not infected with H. pylori remains undefined. Although co-therapy of aspirin with an acid suppressant reduces the risk of ulcer bleeding, drug compliance may limit its clinical usefulness particularly in patients who are already receiving multiple drugs.

ELIGIBILITY:
High risk cohort:

Inclusion Criteria:

1. History of endoscopically confirmed ulcer bleeding
2. Need long-term aspirin for cardiovascular or cerebrovascular prophylaxis
3. A negative test for H. pylori based on histology

Exclusion Criteria:

1. Concomitant use of anti-ulcer drug, anticoagulant, non-aspirin NSAIDs or steroids
2. Current or past H. pylori infection
3. Previous acid-reduction gastric surgery
4. Gastric outlet obstruction, erosive esophagitis, gastroesophageal varices
5. Moribund or incurable cancers

Average-risk cohort

Inclusion criteria:

Patients must fulfill ALL of the following:

1. No history of ulcer bleeding
2. Need long-term aspirin for cardiovascular or cerebrovascular prophylaxis
3. H. pylori positive OR negative

Exclusion criteria:

1. Concomitant use of anti-ulcer drug, anticoagulant, non-aspirin NSAIDs or steroid
2. Previous acid-reduction gastric surgery
3. Moribund or incurable cancers
4. Previous attempts of H. pylori eradication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: High-risk patients were from our hospital while average-risk patients were from our out-patient clinics.
Sampling Method: Non-Probability Sample
Enrollment: 467 (Actual)
Dates: Start 1995-01; Primary Completion 2010-06 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Ulcer complications | 10 years
  defined as bleeding or perforation

CONTACTS AND LOCATIONS:
Overall Officials: Francis KL CHAN, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, China